CLINICAL TRIAL: NCT02757521
Title: Nitrous Oxide - A Novel Therapy for Treatment-Resistant Bipolar Depression
Brief Title: Nitrous TRD Bipolar Depression
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Study sponsor ended trial due to low recruitment
Sponsor: Washington University School of Medicine (Other)
Collaborators: Stanley Medical Research Institute (Other); PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201509128
Record Dates: First submitted 2016-04-14; First posted 2016-05-02 (Estimated); Results first posted 2019-07-05 (Actual); Last update posted 2019-07-05 (Actual); Status verified 2019-04

CONDITIONS: Treatment- Resistant Bipolar Disorder; Bipolar Disorder; Bipolar Depressive Disorder
Keywords: Bipolar Depressive Disorder; Treatment- Resistant Bipolar Disorder; Nitrous Oxide
MeSH Terms: conditions — Bipolar Disorder | interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 50% nitrogen {inert}/ 50% oxygen, 3 one hour inhalation treatments per Stage, every other day (M,W,F)
  Interventions: Drug: Placebo
- Nitrous Oxide (Experimental): 50% nitrous oxide/ 50% oxygen, 3 one hour inhalation treatments per Stage, every other day (M,W,F)
  Interventions: Drug: Nitrous Oxide

INTERVENTIONS:
Drug: Nitrous Oxide — 50% nitrous oxide/ 50% oxygen, 3 one hour inhalation treatments per Stage, every other day (M,W,F)
  Other Names: Laughing Gas
  Arms: Nitrous Oxide
Drug: Placebo — 50% nitrogen {inert}/ 50% oxygen, 3 one hour inhalation treatments per Stage, every other day (M,W,F)
  Arms: Placebo

SUMMARY:
Investigators will study approximately 64 patients with Treatment-Resistant Bipolar Depressive Disorder, defined as a failure of at least 1 antidepressants in the current depressive episode and 2 lifetime medication failures. The study will last approximately 6 to 8 weeks, involving randomization into one of two treatment groups receiving 3 one hour long inhalation treatments over a week.

DETAILED DESCRIPTION:
Investigators will study approximately 64 patients with Treatment-Resistant Bipolar Depressive Disorder, defined as a failure of at least 1 antidepressants in the current depressive episode and 2 lifetime medication failures. The study will last approximately 6 to 8 weeks, involving randomization into one of two treatment groups receiving 3 one hour long inhalation treatments over a week. Post-treatment assessments follow each inhalation treatment and are conducted 1 week and 2 weeks following the final inhalation treatment. Patients are then randomized again into the Second Stage of the study, involving the same treatment and post-treatment schedule as the First Stage detailed above.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18-65 years of age
* Treatment-resistant bipolar depressive disorder without psychosis and a MADRS baseline score of >20. All patients must have history of being on a serum-verified (at time of entry into study) mood stabilizer [lithium at 0.5-1.2mEq/L; or valproic acid, 50-125mcg/ml] for 4 weeks prior to entry into the study and remain on this mood stabilizer during the course of the trial. Further, subjects will have failed two adequate dose/duration antidepressant courses in their lifetime, including one in the current depressive episode (verified by Antidepressant Treatment History Form).
* Good command of the English language

Exclusion Criteria:

* Schizophrenia
* Schizoaffective disorder
* Obsessive-compulsive disorder or panic disorder
* Active or recent substance abuse or dependence (in remission at least 1 year prior to the study; exception = nicotine use disorders)
* A diagnosis of personality disorder that may interfere with the patient's ability to improve on nitrous oxide as determined by study investigator
* Acute medical illness that may pose subject at risk during nitrous oxide administration (neurological disorders or medical disorders including dementia, stroke, encephalopathy, Parkinson's Disease, brain tumors, multiple sclerosis, seizure disorder, severe cardiac disease, any disease known to affect drug metabolism and excretion, i.e. renal or liver disease) per P.I. discretion
* Active suicidal intention (inability to contract for safety)
* Active psychotic symptoms
* Patients with significant pulmonary disease and/or requiring supplemental oxygen
* Contraindication against the use of nitrous oxide: pneumothorax; bowel obstruction; middle ear occlusion; elevated intracranial pressure; chronic cobalamin and/or folate deficiency treated with folic acid or vitamin B12; pregnant patients; breastfeeding women; previous administration of NMDA-receptor antagonists (e.g., ketamine); current electro-convulsive therapy treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-03-25 (Actual); Primary Completion 2016-12-06 (Actual); Study Completion 2016-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Palanca, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Nitrous Oxide
Started | 1 | 0
Completed | 0 | 0
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Population: Difficulty with recruitment caused study sponsor to end trial after designated award length; analysis not done
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nitrous Oxide | Total
Number analyzed (Participants) | 1 | 0 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Full Range); unit: years] | 70 [70 to 70] |  | 70 [70 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 1 |  | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in MADRS (Montgomery Asberg Depression Rating Scale)
Description: Change in depressive symptoms on MADRS scale between baseline and day 7 follow up
Time Frame: up to 1 week
Population: Difficulty with recruitment caused study sponsor to end trial after designated award length; no analysis done
Arm/Group | Placebo | Nitrous Oxide
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Hamilton Depression Rating Scale-17 Item (Ham-D17)
Time Frame: up to1week
Reporting Status: Not Posted

3. Secondary Outcome: Young Mania Rating Scale (YMRS) to Assess Emergence of Mania/Hypomania
Description: Young Mania Rating Scale (YMRS) to assess emergence of mania/hypomania (patients with YMRS scores > 12 will be removed from the trial and recommended for follow up treatment per Psychiatry P.I., i.e., nitrous oxide treatments discontinued)
Time Frame: up to 1 week
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Profile of Mood States (POMS) Short Form to Assess for Rapid/Instantaneous Changes in Mood/Affect
Time Frame: up to 1 week
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Quick Inventory of Depressive Symptomatology- Self Report (QIDS -SR) Patient-rated Depression Measure
Time Frame: up to 1 week
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Clinician Administered Dissociative States Scale (CADSS) for Emergence of Disassociation
Time Frame: up to 1week
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Brief Psychiatric Rating Scale (BPRS) to Assess Psychotic or Hallucinogenic Behavior
Time Frame: up to 1 week
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Scale for Suicidal Ideation (SSI) to Assesses for Emergence of Suicidal Thinking
Time Frame: up to 1 week
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 2 weeks
Description: No participants enrolled in Nitrous Oxide arm
Arm/Group | Placebo | Nitrous Oxide
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=1) | Nitrous Oxide (N=0)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Worsened Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Feeling more cold mostly in feet (General disorders) | 1 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT02757521/Prot_SAP_000.pdf